CLINICAL TRIAL: NCT06706895
Title: A Single-arm, Single-center Phase II Clinical Study on the Clinical Efficacy and Safety of Paclitaxel Polymeric Micelles for Injection Combined With Fruquintinib Capsules in the Second-line Treatment of Patients With Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Director of Oncology Department, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhongshan Hospital
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Advanced Gastric Cancer; Paclitaxel Polymeric Micelles for Injection; Fruquintinib Capsules
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel Polymeric Micelles for Injection combined with Fruquintinib Capsules (Experimental): Fruquintinib Capsules：4 mg / day, orally once daily on days 1-14 in 21-day cycles. If the patient has AE of grade 3 or above, the dose of fruquintinib capsules is reduced to 3 mg / day(dose discontinuation to dose reduction).
  Paclitaxel Polymeric Micelles for Injection：150mg / m2 intravenously over 3 hours on Days1,8 of each 21-day cycle. Do not need special infusion device.
  Paclitaxel Polymeric Micelles for Injection and Fruquintinib Capsules are used for 6 cycles. Subsequently, dual-drug or single-drug maintenance therapy was selected according to the tolerance of the patients. Subsequently, Paclitaxel Polymeric Micelles for Injection ( 120mg / m2, if the patient is intolerable, the dose can be reduced to 100mg / m2 ), until occur the disease progress, the intolerant toxicity or the patient withdrawal.
  Interventions: Drug: Paclitaxel Polymeric Micelles for Injection combined with Fruquintinib Capsules

INTERVENTIONS:
Drug: Paclitaxel Polymeric Micelles for Injection combined with Fruquintinib Capsules — Fruquintinib Capsules：4 mg / day, orally once daily on days 1-14 in 21-day cycles. If the patient has AE of grade 3 or above, the dose of fruquintinib capsules is reduced to 3 mg / day(dose discontinuation to dose reduction).
  Paclitaxel Polymeric Micelles for Injection：150mg / m2 intravenously over 3 hours on Days1,8 of each 21-day cycle. Do not need special infusion device.
  Paclitaxel Polymeric Micelles for Injection and Fruquintinib Capsules are used for 6 cycles. Subsequently, dual-drug or single-drug maintenance therapy was selected according to the tolerance of the patients. Subsequently, Paclitaxel Polymeric Micelles for Injection ( 120mg / m2, if the patient is intolerable, the dose can be reduced to 100mg / m2 ), until occur the disease progress, the intolerant toxicity or the patient withdrawal.

SUMMARY:
This study is a single-arm, open, phase II clinical trial aimed at evaluating the anti-tumor efficacy and safety of paclitaxel polymeric micelles for injection combined with furquintinib as second-line treatment for advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

- 1.Age ≥ 18 years ; 2. Histologically confirmed advanced gastric cancer. The first-line systemic treatment containing oxaliplatin and fluorouracil failed. According to RECIST version 1.1, there is at least one measurable lesion; 3. Eastern Cooperative Oncology Group（ECOG）score 0 or 1 ; 4.Expected survival ≥ 12 weeks ; 5.Adequate organ and bone marrow function (no hematopoietic growth factor, blood transfusion or platelet therapy was given within 1 week before the first drug treatment ):

1. Blood routine: leucocyte ≥3.0×109/L, absolute neutrophil count (ANC)≥1.5 ×109/L, platelet count（PLT）≥ 100×109/L, Hemoglobin ( Hb )≥ 9.0 g/dL;
2. Liver function : total bilirubin ≤ 1.5 ×ULN;Alanine aminotransferase(ALT)/aspartate aminotransferase (AST)≤2.5×ULN without liver metastasis ;ALT/AST ≤ 5 ×ULN with liver metastasis;
3. Coagulation function : international normalized ratio (INR)≤1.5×ULN, and activated partial thromboplastin time (APTT) ≤1.5×ULN ;(Investigator judge that INR and APTT should be in the safe and effective treatment range for patients who are undergoing anticoagulant therapy);
4. Renal function : serum creatinine ≤ 1.5×ULN ;
5. Adequate cardiac function, left ventricular ejection fraction (LVEF) > 50 % detected by two-dimensional echocardiography.

6.Understand the research and voluntarily sign the informed consent.

Exclusion Criteria:

* 1. Patients have received clinical trials of other research drugs or research instruments within 28 days before the first study of treatment ;or received anti-tumor treatment including but not limited chemotherapy, radiotherapy (excluding palliative radiotherapy completed at least 1 week before the treatment )and targeted therapy within 2 weeks before the first study of treatment; 2.The toxicity of previous anti-tumor therapy has not returned to the level of 0 or 1 (excluding alopecia ， peripheral neurotoxicity caused by chemotherapy ≤ 2) ; 3.Surgery was performed within 4 weeks before the first treatment (except biopsy) or the surgical incision was not completely healed ; 4. There were ascites requiring drainage or diuretic treatment, or pleural effusion or pericardial effusion requiring drainage or accompanied by shortness of breath within 2 weeks before the first treatment; 5.Symptomatic brain metastasis or spinal cord compression(except for previously treated patients with brain metastases, if the clinical condition was stable within 4 weeks before the first treatment and the imaging evidence did not show disease progression).

  6. History of other primary malignant tumors in the past 5 years (except for malignant tumors that have been cured, e,g, basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in situ, breast cancer in situ).

  7.History of HIV, or active bacterial or fungal infection requiring systematic treatment within 14 days before the first treatment .

  8. HBV DNA ≥ 104copies / ml or > 2000IU / ml in the screening period ; 9.Cardiovascular diseases with significant clinical significance, including but not limited acute myocardial infarction, severe / unstable angina, cerebrovascular accident or transient ischemic attack, congestive heart failure (New York Heart Association classification > 2) within 6 months before enrollment;other arrhythmia treated with drugs(exclude β blockers or digoxin); electrocardiogram repeated detection of QTcF interval ≥ 450 ms.; hypertension failed to be well controlled after antihypertensive drug treatment (systolic blood pressure > 150 mmHg, diastolic blood pressure > 100 mmHg ).

  10.Clinically significant abnormalities in serum electrolyte levels ; 11.Women during pregnancy or lactation ; 12.Fertile but unwilling to accept effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 24 months
  PFS(Progression-Free-Survival) was the time from randomization until the date of objectively determined progressive disease (PD) or death due to any cause, whichever occurred first.